CLINICAL TRIAL: NCT03156257
Title: OR-DRPD-SRI/CASIS2016: The Role of the Space Environment on Vascular Endothelial and Smooth Muscle Cell Processes
Brief Title: The Role of the Space Environment on Vascular Endothelial and Smooth Muscle Cell Processes
Acronym: OR-DRPD-SRI
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Florida Space Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB201700080; P0036354 (Other Grant/Funding Number: Florida Space Institute)
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cardiovascular Diseases
Keywords: Microgravity Effects on Vascular Cells
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Self-reported healthy males and females: The investigators are interested in sampling a wide variety of individuals from varying ethnic groups, sex, and age range.
  Interventions: Biological: Blood volume collected specifically for this study

INTERVENTIONS:
Biological: Blood volume collected specifically for this study — The subject will be sitting in a chair, and a needle will be inserted into a vein in their arm. Study Team will draw about 45ml or 3 tablespoons of whole blood for research.

SUMMARY:
By studying the affect of the space environment on vascular cell types, our goal is to elucidate the mechanism of vascular cell damage in the space environment by exposing vascular cells to space flight. In this pilot study, The study team propose to assess changes in transcriptomics of vascular cell types in space compared to those in a ground based study.

DETAILED DESCRIPTION:
Under conditions of simulated microgravity, it is well known that normal cellular processes of vascular cells are altered. While these studies provide important information about these alterations in cells, it is likely not a complete picture due to the limitations of ground based simulated microgravity. It is our hypothesis that real microgravity, as is experienced in space, will reveal changes in EC and SMC phenotype and function that alters cell-cell communication. The study team will test our hypothesis by culturing mature endothelial cells, as well as stem cell derived endothelial cells, and mature smooth muscle cells in low Earth orbit (LEO) on the International Space Station (ISS) U.S. National Laboratory. The specific aims the Study team have proposed are the following:

Specific Aim #1: Preflight isolation and characterization of circulating stem cell derived endothelial cells. Specifically, the Study team will isolate CSCs from whole blood then direct them down an EC pathway. Once differentiated the study team will characterize their phenotype.

Specific Aim #2: Culture mature ECs, SMCs, and CSC derived ECs under conditions of low Earth orbit (LEO) aboard the ISS. Specifically, The study team will use advanced flight hardware to establish an active cell culture on the ISS. The cells will be cultured for a duration of 3 and 10 days, at which time the cells will be frozen for subsequent analysis. Simultaneously, the study team will culture the same populations in a ground based microgravity simulator as well as a normal gravity control.

Specific Aim #3: Assess the morphologic and genetic changes in cells after 3 and 10 days of space flight. Specifically, upon return to Earth, a transcriptome analysis will be completed from the frozen cell samples to assess changes in the cells molecular machinery.

This proposed study builds upon the abundant literature, including our own, surrounding the effects of ground based simulated microgravity on vascular endothelial cells. However, the study team include the less studied populations of smooth muscle cells and stem cell derived ECs. The goal of this work is to leverage conditions on the ISS, a powerful one-of-a-kind microgravity research platform in low Earth orbit, to study these cells and their cellular processes as it relates to cardiovascular disease (CVD) and cardiovascular deconditioning. This work seeks to reveal currently unknown changes in vascular cell health that lead to these diseases. The impact of this work is broad and can lead to new treatment options for millions of people who suffer from CVD including neointimal hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported healthy individuals
* Willingness to have 50mls of whole blood collected

Exclusion Criteria:

* Unwillingness to have blood used in stem cell research

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The Study team is interested in sampling a wide variety of health individuals from varying ethnic groups, sex, and age range.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Changes in gene expression in space vs earth cultured vascular cells | within 1 year of collecting cells
  Post space flight the study team will conduct transcriptomics analysis to assess changes in the cells grown in space (microgravity), on earth (normal gravity), and in a rotating wall vessel bioreactor (ground based simulated microgravity)

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Allen, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided